CLINICAL TRIAL: NCT05863481
Title: Obstetric Outcome in Pregnancies Treated With Laparoscopic Cerclage: an Observational Study in a Danish Cohort
Brief Title: Obstetric Outcome in Pregnancies Treated With Laparoscopic Cerclage
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: LapAUH
Record Dates: First submitted 2023-05-04; First posted 2023-05-18 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-05

CONDITIONS: Pre-Term; Cervical Insufficiency
MeSH Terms: conditions — Premature Birth; Uterine Cervical Incompetence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopic cerclage: Patients who underwent laparoscopic cerclage at Aarhus University Hospital, Denmark in the study period
  Interventions: Procedure: Laparoscopic cerclage placement

INTERVENTIONS:
Procedure: Laparoscopic cerclage placement — The surgical method of the laparoscopic cerclage procedure at Aarhus University Hospital previous described in a paper by Riiskjaer et al (DOI: 10.1111/aogs.12001)

SUMMARY:
Preterm birth is a leading cause of neonatal mortality and morbidity. Cervical insufficiency is one factor implicated in the complex mechanisms involved in spontaneous preterm birth. Trans-abdominal insertion of a cervical cerclage suture can be used to treat cervical insufficiency. Growing evidence support that laparoscopic cerclage procedures are safe and effective. Still, many aspects of the laparoscopic cerclage remains uncertain. Therefore, the investigators plan to study the obstetric outcome from the first and subsequent pregnancies after laparoscopic cerclage in a Danish cohort from Aarhus University Hospital in a 10 years' period.

DETAILED DESCRIPTION:
Please see attached study protocol for further desricption.

ELIGIBILITY:
Inclusion Criteria:

* Persons who underwent laparoscopic cerclage at Aarhus University Hospital, Denmark between May 2011 and May 2021

Exclusion Criteria:

* Persons who had their laparoscopic cerclage performed subsequently to a trachelectomy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons at risk of preterm birth who were offered and underwent laparoscopic cerclage surgery at Aarhus University Hospital, Denmark in the period from May 2011 till May 2021.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Neonatal survival (defined as survival at time of discharge from hospital) | From birth until discharge, an average of 8 weeks
  no. (reported for first, and consecutive deliveries)

SECONDARY OUTCOMES:
Number of neonates surviving with major neonatal morbidity | From birth until discharge, an average of 8 weeks
  * Necrotising enterocolitis (NEC) (no.)
  * Bronchopulmonary Dysplasia (BPD) (defined as respiratory/oxygen support at postmenstrual age (PMA) 36 weeks) (no.)
  * Intraventricular haemorrhage (IVH) Grade III and IV (no.)
  * Hydrocephalus with ventriculoperitoneal (VP) shunt (no.)
  * Periventricular leukomalacia (no.)
  * Retinopathy of prematurity (ROP) (no.) (Reported for first, and consecutive deliveries)
Number of pregnancies | From the laparoscopic cerclage until May 1, 2023 (two years after the enrollment period ends)
  no.
Number of miscarriages | From the laparoscopic cerclage until May 1, 2023 (two years after the enrollment period ends)
  * Early miscarriages (<16 weeks and 0 days) (no.)
  * Late miscarriages (<22 weeks and 0 days) (no.)
Deliveries | From birth until discharge, an average of 8 weeks
  * Deliveries <28 weeks and 0 days of an infant living (no.)
  * Deliveries <32 weeks and 0 days of an infant living (no.)
  * Deliveries <34 weeks and 0 days of an infant living (no.)
  * Deliveries <37 weeks and 0 days of an infant living (no.) (reported for first, and consecutive deliveries)
Number of uterine ruptures | From the laparoscopic cerclage until May 1, 2023 (two years after the enrollment period ends)
  no.
Time to first pregnancy (years and days) | From the laparoscopic cerclage until May 1, 2023 (two years after the enrollment period ends)
  no.

OTHER OUTCOMES:
Neonatal characteristics | At delivery
  * Gestational age (weeks and days) (no.)
  * Birthweight (grams) (Reported for deliveries with a gestational age ≥ 20 weeks and 0 days - allow missing data)
Number of early complications from the laparoscopic cerclage procedure | 30 days from the procedure
  * Conversion to laparotomy during surgery (no.)
  * Haemorrhage > 500 ml (no.)
  * Postoperative infection treated at hospital (no.)
  * Damage to internal organs (no.)
  * Need for re-operation (no.)
  * Admission to Intensive Care Unit (no.)
  * Thromboembolic events (defined as deep vein thrombosis, pulmonary embolism or stroke) (no.)
  * Maternal cardiopulmonary arrest (no.)
  * Maternal death (no.)
Number of late complications from the laparoscopic cerclage procedure | From the laparoscopic cerclage until May 1, 2023 (two years after the enrollment period ends)
  * Erosion into the vagina treated in hospital (no.)
  * Pain complaints from the stiches leading to intervention in pregnancy (no.)
  * Other complications from the cerclage leading to intervention in hospital (no.)

CONTACTS AND LOCATIONS:
Overall Officials: Lise Q Krogh, MD, Principal Investigator — Aarhus University Hospital/Aarhus University

DOCUMENTS (2):
  • Study Protocol (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT05863481/Prot_003.pdf
  • Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT05863481/SAP_004.pdf